CLINICAL TRIAL: NCT05880121
Title: Neuron-specific Humoral and Cellular Immune Correlates of Structural and Functional Brain Connectomics in Neuropsychiatric Lupus
Acronym: INLES
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Giuseppe A. Ramirez, Dr., IRCCS San Raffaele
Other Study IDs: GR-2021-12372172
Record Dates: First submitted 2023-05-05; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- systemic lupus erythematosus: Patients with SLE according to the 1997 ACR, 2012 SLICC or 2019 EULAR/ACR criteria will undergo MRI along with neuropsychological tests, rheumatological evaluation and blood sample collection at baseline and after at least 12 months or during a new neuropsychiatric manifestation. In case of existing MRI with compatible features, they will be used as baseline studies.
  Interventions: Diagnostic Test: MRI
- healthy controls: Subjects with Charlson's Comorbidity Index=0 with no ongoing chronic therapy and no history of immune-mediated disease will undergo a single MRI study, along with neuropsychological tests and blood sample collection. In case of existing MRI with compatible features, no additional studies will be performed in this cohort.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — brain MRI

SUMMARY:
Systemic lupus erythematosus (SLE) is the prototype systemic autoimmune disease. Neuropsychiatric SLE (NPSLE) is a major cause of morbidity. Its pathophysiology remains unclear and target autoantigens have not yet been identified. Site- specific autoantigen expression might correlate with imaging abnormalities. Based on existing expertise on the use of peptide/protein arrays and on antigen-specific T cell tracking, we plan to identify new fingerprints and targets for NPSLE. SLE patients +/- NPSLE and healthy subjects will undergo advanced magnetic resonance imaging. Three-dimensional data on structural or functional brain architecture will be integrated with brain transcriptome atlases and candidate antigens for autoreactive autoantibodies and T lymphocytes identified and validated. The evidence will add to current knowledge on NPSLE pathophysiology, provide new multimodal diagnostic tools for better patient care and a platform for innovative, personalized treatments.

ELIGIBILITY:
Inclusion Criteria:

Patients with SLE

* Diagnosis of SLE according to the ACR 1997, SLICC 2012 or EULAR/ACR 2019 criteria
* age ≥ 18 years (reference centre)
* age 15-17 years (affiliated centre)

Healthy subjects

* Charlson's Comorbidity Index=0 and no chronic treatment
* age ≥ 18 years (reference centre)
* age 15-17 years (affiliated centre)

Exclusion Criteria:

* History of T-cell neoplasia
* Active B-cell neoplasia or history of B-cell neoplasia of less than five years
* Contraindications to MRI
* Pregnancy
* Ongoing or past treatment with T-depleting agents
* History of brain cancer
* History of congenital brain disorders
* Cerebral disorders secondary to trauma, toxins or other metabolic or environmental factors unrelated to SLE according to the Investigator's evaluation
* Any other condition conferring excessive physical and psychological risk to the subject according to the Investigator's opinion

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: see above
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
To detect regional brain functional abnormalities in patients with SLE through advanced magnetic resonance imaging (MRI). | 12 months (extensions allowed for existing images before study onset)
  All study subjects will be assessed at baseline through 3T MRI. Repeat MRI will be performed after at least 12 months or in case of new neuropsychiatric events in all patients with SLE. The MRI protocol will include conventional structural sequences (3D fluid-attenuated inversion recovery [FLAIR], 3D T1-weighted inversion recovery prepared gradient echo), advanced structural sequences (diffusion-weighted [DW] pulsed-gradient spin-echo [PSGE] single-shot echo-planar imaging, optimized for an accurate estimation of the neuriteorientation dispersion and density imaging [NODDI] model), and functional MRI sequences acquired in resting-state condition.
To identify autoantigen-specific circulating antibodies associated with neuropsychiatric morbidity and imaging features in patients with SLE. | 12 months (extensions allowed for existing MRI images before study onset)
  High-throughput peptide and/or protein arrays customised according to the data derived from neuroimaging-annotated transcriptome analyses and/or from previous evidence from immune studies performed in a large multicentre cohort of patients with SLE (ZEUS study: NCT02403115) will be used to define candidate antigen targets for autoantibodies. Serum samples will be collected longitudinally at time of clinical evaluation and neuroimaging and analysed by ELISA.
To correlate antigen-specific CD4+ T-cell dynamics over time with the spectrum of SLE, NPSLE and associated MRI findings. | 12 months (extensions allowed for existing MRI images before study onset)
  Major histocompatibility complex (MHC) multimers bound to relevant autoepitopes identified through in silico analyses of data from neuroimaging-annotated transcriptome analyses and/or from previous evidence from immune studies performed in a large multicentre cohort of patients with SLE (ZEUS study: NCT02403115) will be used to detect and track antigen-specific CD4+ T-cells. Further characterisation of T-cells will be performed in terms of differentiation and polarisation. In vitro T-cell reactivity assays with relevant autoepitopes will also be performed

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided